CLINICAL TRIAL: NCT02948985
Title: Evaluation of Individual Peripheral Blood Circulating Tumor Cells Combined With Tumor Marker Detection of Efficacy of Chemotherapy in Patients With Advanced Colorectal Cancer: A Observational Clinical Trial
Brief Title: Evaluation of CTCs Combined With Tumor Marker Detection of Efficacy of Chemotherapy in mCRC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qi Li, Executive director of cancer center, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Shanghai1stQli01
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Metastatic colorectal cancer; Cetuximab; CTCs; ct DNA
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Peripheral blood samples of 10 mL were collected from the patients for ctDNA and CTCs analysis

GROUPS / COHORTS (1):
- RAS and B-raf wild type mCRC: patients with histologically confirmed RAS and B-raf wild type mCRC treated with FOLFIRI±cetuximab
  Interventions: Other: treated with FOLFIRI±cetuximab

INTERVENTIONS:
Other: treated with FOLFIRI±cetuximab — Peripheral blood samples of 10 mL were collected from the patients for CTCs analysis and tumor marker in every cycle D0 and D8. Tumor response evaluation will be performed after four cycles of chemotherapy by CT/MRI based on RECIST. Clinical data, including tumor stage, metastatic organ, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.The correlation of the RAS status on CTCs and the mutant gene in ctDNA to the therapeutic response will be evaluated.

SUMMARY:
Evaluation of individual peripheral blood circulating tumor cells combined with tumor marker detection of efficacy of chemotherapy in patients with advanced colorectal cancer: A observational clinical trial

DETAILED DESCRIPTION:
In 2004, based on AVF2107g clinical research, FDA has approved bevacizumab as first targeted drugs for the treatment of advanced colorectal cancer[1].So far, chemotherapy combined with target agents is currently first line standard of patients with advanced colorectal cancer. The anti-EGFR monoclonal antibodies((cetuximab and panitumumab) also have been demonstrated to be efficient in the treatment of metastatic colorectal cancer. In the CRYSTAL and OPUS studies, adding cetuximab to first-line chemotherapy (CT) improved clinical benefit in patients (pts) with KRAS wild-type (wt) mCRC [2,3]. FIRE-3 and TAILOR once again proved cetuximab combined FORFIRI or FOLFOX will improved clinical benefit[4]. Target agents are expensive, so It is necessary to explore a new evaluation criteria to avoid unnecessary economic waste.

RECIST(Response Evaluation Criteria in Solid Tumors) is not suitable for the target or immunotherapy. The effect of chemotherapy not only displayed as morphology(tumor size reduction), but also as the biological activity change of tumor cells(e.g.cystic degeneration and cavity).PET-CT combined imaging of molecular function and morphology, but PET-CT was low cost -effective. The tumor markers is a rapid, easy to repeat method, but the change of the markers can not evaluation the response of tumor as an individual indicator. So we need a more sensitive effective evaluation marker.

Circulating tumor cells (CTCs) are rare cancer cells released from tumors into the bloodstream that are thought to have a key role in cancer metastasis. The distant metastasis is the leading cause of death in patients with mCRC. CTCs is a method to detect the early tumor micrometastasis. CTCs is predictive of PFS and OS in lung cancer and breast cancer. CTCs is also predictive of response of tumor. CTCs is more accuracy, more sensitive way than imageology or other tumor marker to predict therapy effect and outcome.

The anti-EGFR monoclonal antibody (cetuximab) target the human epidermal growth factor receptor and have been integrated into treatment regimens of mCRC. The EGFR expression is not the predicted marker of cetuximab, in patients who express EGFR, the ORR only 10%-20%[5,6].In CRYSTAL, The addition of cetuximab to FOLFIRI as first-line therapy improves PFS in patients with KRASwild-type mCRC[2]. Up to now, we know only RAS wild type patients would benefit from anti-EGFR therapy.[7] The CALGB/SWOG80405 confirmed the conclusion. Some study also found the patients with B-raf (V600e) mutation would not benefit from anti-EGFR therapy[8]. Taken together, we need a more accuracy, more sensitive method to predict the effect of cetuximab.

The study is a single arm, single-center, observational study undertaken in anticipated 100 patients with histologically confirmed RAS and B-raf wild type mCRC. These patients received FOLFIRI±cetuximab therapy.

Peripheral blood samples of 10 mL were collected from the patients for CTCs analysis and tumor marker in every cycle D0 and D8. The CTCs sued the integrated subtraction enrichment (SET) and immunostaining-fluorescence in situ hybridization (iFISH) platform.Tumor assessments will be performed every four cycles based on RECIST v1.1 criteria using CT/MRI scan. If the assessments are inconsistent, we will collect 10ml peripheral blood for ct DNA test, which using BEAMing, to analyze mutant gene.

The correlation of the RAS status on CTCs and the mutant gene in ctDNA to the therapeutic response will be evaluated, and found the cut-off of CTCs.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age18-75 years old
* Histologically confirmed mCRC
* First metastatic,unresectable
* RAS and B-raf wild type
* .At least one measurable disease according to the RECIST criteria by CT/MRI
* Expected survival time≥12 weeks
* ECOG PS 0-1
* Adequate bone marrow, hepatic, renal and metabolic function

Exclusion Criteria:

* Received chemotherapy for CRC previously, except adjuvant chemotherapy end of adjuvant chemotherapy≥9m(contain irinotecan) or ≥9m(not contain irinotecan) before the study.
* Surgery or radiotherapy ≤30 days before the study.
* Received anti-EGFR,anti-VEGF or other signaling pathway inhibitor previously

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed RAS and B-raf wild type mCRC treated withFOLFIRI±cetuximab
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of RAS status on CTCs with clinical outcomes | 3 years
  To evaluate the correlation of CTCs and their RAS status to the clinical outcomes

SECONDARY OUTCOMES:
Correlation of mutant gene in ctDNA with cetuximab resistance. | 3 years
  To evaluate the correlation of mutant gene in ctDNA to the cetuximab resistance

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xingpeng, MD PHD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine

REFERENCES:
- [Result] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Result] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720
- [Result] Bokemeyer C, Van Cutsem E, Rougier P, Ciardiello F, Heeger S, Schlichting M, Celik I, Kohne CH. Addition of cetuximab to chemotherapy as first-line treatment for KRAS wild-type metastatic colorectal cancer: pooled analysis of the CRYSTAL and OPUS randomised clinical trials. Eur J Cancer. 2012 Jul;48(10):1466-75. doi: 10.1016/j.ejca.2012.02.057. Epub 2012 Mar 23. PMID 22446022
- [Result] Heinemann V, von Weikersthal LF, Decker T, Kiani A, Vehling-Kaiser U, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Hielscher J, Scholz M, Muller S, Link H, Niederle N, Rost A, Hoffkes HG, Moehler M, Lindig RU, Modest DP, Rossius L, Kirchner T, Jung A, Stintzing S. FOLFIRI plus cetuximab versus FOLFIRI plus bevacizumab as first-line treatment for patients with metastatic colorectal cancer (FIRE-3): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Sep;15(10):1065-75. doi: 10.1016/S1470-2045(14)70330-4. Epub 2014 Jul 31. PMID 25088940
- [Result] Cunningham D, Humblet Y, Siena S, Khayat D, Bleiberg H, Santoro A, Bets D, Mueser M, Harstrick A, Verslype C, Chau I, Van Cutsem E. Cetuximab monotherapy and cetuximab plus irinotecan in irinotecan-refractory metastatic colorectal cancer. N Engl J Med. 2004 Jul 22;351(4):337-45. doi: 10.1056/NEJMoa033025. PMID 15269313
- [Result] Saltz LB, Meropol NJ, Loehrer PJ Sr, Needle MN, Kopit J, Mayer RJ. Phase II trial of cetuximab in patients with refractory colorectal cancer that expresses the epidermal growth factor receptor. J Clin Oncol. 2004 Apr 1;22(7):1201-8. doi: 10.1200/JCO.2004.10.182. Epub 2004 Mar 1. PMID 14993230
- [Result] Sorich MJ, Wiese MD, Rowland A, Kichenadasse G, McKinnon RA, Karapetis CS. Extended RAS mutations and anti-EGFR monoclonal antibody survival benefit in metastatic colorectal cancer: a meta-analysis of randomized, controlled trials. Ann Oncol. 2015 Jan;26(1):13-21. doi: 10.1093/annonc/mdu378. Epub 2014 Aug 12. PMID 25115304
- [Result] Tol J, Nagtegaal ID, Punt CJ. BRAF mutation in metastatic colorectal cancer. N Engl J Med. 2009 Jul 2;361(1):98-9. doi: 10.1056/NEJMc0904160. No abstract available. PMID 19571295